CLINICAL TRIAL: NCT02976610
Title: Open Label, Single Center Clinical Trial of a Novel Hemolysis Point of Care Test at an Emergency Department.
Brief Title: Clinical Study of a Novel Hemolysis Point of Care Test at an Emergency Department.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hemcheck Sweden AB (Industry)
Collaborators: Landstinget i Värmland (Other)
Responsible Party: Principal Investigator, Lars-Olof Hansson, Clinical chemist, physician., Landstinget i Värmland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HC001
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Hemolysis; Blood Specimen Collection
Keywords: hemolysis
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): This is the control group where no intervention takes place. Blood sampling carried out according to routine at the emergency department.
- 2 (Experimental): During the blood sampling the health care professional will screen all vacuum Lithium Heparin tubes, with the Hemolysis point-of-care test (H-POCT). If the health care professional receives a negative test the bloodsample is sent to the local laboratory.
  If H-POCT indicates a positive test, of free hemoglobin in plasma, the bloodsample and H-POCT will be discarded and a new sample will be collected and screened for hemolysis. This can be repeated 3 times.
  Interventions: Device: Hemolysis Point-of-Care test

INTERVENTIONS:
Device: Hemolysis Point-of-Care test — Hemolysis measurement of plasma using a point of care test to determine the hemolysis level in plasma
  Arms: 2

SUMMARY:
This study aims to investigate the outcome of hemolysis frequency when a hemolysis point of care test is introduced in an emergency department.

DETAILED DESCRIPTION:
In a blood sample process, the preanalytical phase is accountable for a vast majority of laboratory test errors. Among preanalytical errors, hemolysis is the most frequent error of sample rejection. Recollection of blood from the patient causes extra suffering, increased turn-around-time hence delayed treatment, and unnecessary extra costs for the health care system.

Here is a novel method for hemolysis point of care detection (H-POCT) evaluated. The single use test is attached to the blood sample in direct conjunction to the sampling process.

Patients will be selected by consecutive selection at the emergency department if blood tests ordered by the physician meet the inclusion criteria. Patients will be randomized into one of two groups. All health care professionals participating in this study has attended in a standard education program in operating H-POCT.

If Allocated into the control group, n: 750, nurses and enrolled nurses will perform blood sample according to routine.

If allocated into the intervention group, n: 750, nurses and enrolled nurses will perform blood sample according to routine and screen all Lithium Heparin vacuum tubes. (for one or all of the analyzes: Liver status, Electrolytes and Troponin T.)

If the hemolysis point of care test (H-poct) indicate a positive test result the Lithium Heparin vacuum tube and the attached H-poct will be discarded and a new sample will be collected and screened for hemolysis until the user receives a negative sample that is not hemolyzed.

This study takes place in a county hospital with 430 beds and the emergency department treats 59000 patients yearly.

ELIGIBILITY:
Inclusion Criteria:

Blood sample analysis ordered:

* Electrolyte
* Troponin T
* ALAT, ASAT, ALP.

Exclusion Criteria:

* Incompletely filled tubes
* Minors (< 18 years)
* Patient not fit according to the health care professional assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1671 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Hemolysis frequency. | Through 52 weeks
  Compare the volume of hemolyzed blood samples in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Hansson, MD-PhD, Study Chair — Landstinget i Värmland; Anders Hallberg, MD-PhD, Study Chair — Centrum för klinisk forskning, SCK, Älvgatan 49, 651 85 Karlstad
Locations (1):
- Emergency department, Central Hospital Karlstad, Karlstad, Värmland County, Sweden

IPD SHARING:
Plan to Share IPD: No